CLINICAL TRIAL: NCT03682185
Title: The Role of Palliative Care Interventions to Reduce Circadian Rhythm Disorders in Persons With Dementia: The Healthy Patterns Study
Brief Title: The Healthy Patterns Sleep Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 825000; 1R01NR015226-01A1 (NIH)
Record Dates: First submitted 2018-04-09; First posted 2018-09-24 (Actual); Results first posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Dementia; Alzheimer Disease; Circadian Rhythm Disorders; Circadian Rhythm Sleep Disorder; Insomnia; Hypersomnia; Cognitive Impairment; Cognitive Decline; Mild Cognitive Impairment; Frontotemporal Dementia; Neurocognitive Disorders; Vascular Dementia; Sleep Disorder; Memory Impairment
Keywords: Neuropsychiatric Behaviors; Agitation; Alzheimer's Disease; Dementia
MeSH Terms: conditions — Dementia; Alzheimer Disease; Chronobiology Disorders; Sleep Disorders, Circadian Rhythm; Sleep Initiation and Maintenance Disorders; Disorders of Excessive Somnolence; Cognitive Dysfunction; Frontotemporal Dementia; Neurocognitive Disorders; Dementia, Vascular; Sleep Wake Disorders; Memory Disorders; Psychomotor Agitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Timed Activity Intervention Protocol (Experimental): The timed activity group will involve 4 in-home visits and 4 brief telephone education sessions provided over 4 weeks. The timed activity intervention provides activities delivered at specific times in the daily cycle. The in-home sessions are spaced weekly so that the participants can have the opportunity to practice the activity with the interventionist and then on their own. During each session, the interventionist will reinforce activity use, review problem solving approaches, and provide education.
  Interventions: Behavioral: Timed Activity Intervention
- Attention-Control Condition (Active Comparator): This condition will contain no active elements beyond its nonspecific components, and no theoretical basis to support an effect on CRDs. The attention-control group will also involve 4 in-home visits and 4 brief telephone education sessions. The attention control group will receive printed educational and training materials from the Alzheimer's Association and the NIH on home modification, health promotion, talking to your doctor, and advanced care planning that coincide with session content.
  Interventions: Behavioral: Attention-Control Condition

INTERVENTIONS:
Behavioral: Attention-Control Condition — This condition will contain no active elements beyond its nonspecific components, and no theoretical basis to support an effect on CRDs. The attention-control group will also involve 4 in-home visits and 4 brief telephone education sessions. The attention control group will receive printed educational and training materials from the Alzheimer's Association and the NIH on home modification, health promotion, talking to your doctor, and advanced care planning that coincide with session content.
  Arms: Attention-Control Condition
Behavioral: Timed Activity Intervention — The timed activity group will involve 4 in-home visits and 4 brief telephone education sessions provided over 4 weeks. The timed activity intervention provides activities delivered at specific times in the daily cycle. The in-home sessions are spaced weekly so that the participants can have the opportunity to practice the activity with the interventionist and then on their own. During each session, the interventionist will reinforce activity use, review problem-solving approaches, and provide education.
  Arms: Timed Activity Intervention Protocol

SUMMARY:
The Healthy Patterns Study intervention is a home-based activity intervention designed to improve symptoms of circadian rhythm disorders (CRD) and quality of life (QOL) in home-dwelling persons with dementia. We will use a randomized two-group parallel design of 200 people with dementia and their caregivers assigned to intervention or attention control groups.

DETAILED DESCRIPTION:
Over 5 million Americans have Alzheimer's disease or a related dementia, a progressive and fatal neurodegenerative condition, affecting close to 15 million family caregivers (CG). Circadian rhythm disorders (CRDs) occur in the majority of persons with dementia and include late afternoon/evening agitation (e.g. sundowning) and irregular sleep-wake rhythms such as daytime hypersomnia, frequent night awakenings, and poor sleep efficiency. CRDs can cause a specific cluster of neuropsychiatric symptoms that occur in over 60 percent of patients with dementia and are associated with increased morbidity and mortality and decreased quality of life. Regulating the circadian system via different types of activity have been shown to alter core clock processes that drive CRD symptoms and suggests that a combination of cognitive, physical, and sensory-based activities, delivered at strategic times, may be an effective mechanism to reduce neuropsychiatric symptoms, decrease sleep disruptions, and enhance quality of life for both the care receiver and the caregiver.

Specific components of this brief, one-month, eight sessions, home-based intervention include: 1) assessing PWD health/functional status and preferences/interests; 2) educating caregivers on environmental cues to promote activity and sleep; and 3) training of caregivers in using timed morning, afternoon, and evening activities based on circadian needs across the day.

ELIGIBILITY:
Inclusion criteria for care receiver (CR):

1. be over age 60
2. English speaking
3. be able to tolerate wrist actigraphy (wear a watch on their wrist for a month)
4. diagnosed with dementia using standard assessments and diagnostic criteria
5. has CG reporting the presence of CRD symptoms
6. If the CR is on any of four classes of psychotropic medications (antidepressant, benzodiazepines, antipsychotic, or anti-convulsant) or an anti-dementia medication (memantine or a cholinesterase inhibitor), we will require that the CR have been on a stable dose for 90 days prior to enrollment (typical time frame in clinical trials) to minimize possible confounding effects of concomitant medications

Inclusion criteria for caregiver (CG):

1. CG is at least 18 years old
2. CG lives close to the participant
3. CG is planning to live in the area for at least 6 months
4. If CG is on a psychotropic medication, CG must be on a stable dose for at least 60 days

Exclusion criteria for CR:

1. deemed to be in a crisis/unsafe situation at baseline
2. reported planned transition to another residential or care setting in less than 6 months
3. at end-stage disease (defined as bed-bound and noncommunicative, or on hospice at baseline)
4. currently enrolled in an interventional clinical trial for dementia or associated symptoms
5. regular use of medications with substantial known effects on the measurement of HPA activity (e.g. corticosteroids, interferons, beta-blockers, cytotoxic chemotherapy)
6. major surgery in the past 3 months
7. history of major psychiatric and/or personality disorder
8. history of heavy cigarette smoking (e.g. than 50 pack years)
9. loss of a loved one in the past 3 months
10. conditions known to affect measurement of circadian rhythm such as use of sedatives/ hypnotics, Huntington's disease, Cushing's disease, Addison's disease, normal pressure hydrocephalus, Parkinson's disease, advanced heart failure (New York Heart Stage 3-4), morbid obesity (BMI 35)

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A. Hodgson, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hodgson NA, Granger DA. Collecting saliva and measuring salivary cortisol and alpha-amylase in frail community residing older adults via family caregivers. J Vis Exp. 2013 Dec 18;(82):e50815. doi: 10.3791/50815. PMID 24378361
- [Background] Hodgson NA, Gitlin LN, Winter L, Czekanski K. Undiagnosed illness and neuropsychiatric behaviors in community residing older adults with dementia. Alzheimer Dis Assoc Disord. 2011 Apr-Jun;25(2):109-15. doi: 10.1097/WAD.0b013e3181f8520a. PMID 20921879
- [Background] Hodgson NA, Andersen S. The clinical efficacy of reflexology in nursing home residents with dementia. J Altern Complement Med. 2008 Apr;14(3):269-75. doi: 10.1089/acm.2007.0577. PMID 18370580
- [Background] Hirschman KB, Hodgson NA. Evidence-Based Interventions for Transitions in Care for Individuals Living With Dementia. Gerontologist. 2018 Jan 18;58(suppl_1):S129-S140. doi: 10.1093/geront/gnx152. PMID 29361067
- [Background] Samus QM, Black BS, Bovenkamp D, Buckley M, Callahan C, Davis K, Gitlin LN, Hodgson N, Johnston D, Kales HC, Karel M, Kenney JJ, Ling SM, Panchal M, Reuland M, Willink A, Lyketsos CG. Home is where the future is: The BrightFocus Foundation consensus panel on dementia care. Alzheimers Dement. 2018 Jan;14(1):104-114. doi: 10.1016/j.jalz.2017.10.006. Epub 2017 Nov 21. PMID 29161539
- [Background] Regier NG, Hodgson NA, Gitlin LN. Characteristics of Activities for Persons With Dementia at the Mild, Moderate, and Severe Stages. Gerontologist. 2017 Oct 1;57(5):987-997. doi: 10.1093/geront/gnw133. PMID 27986794
- [Background] Gitlin LN, Piersol CV, Hodgson N, Marx K, Roth DL, Johnston D, Samus Q, Pizzi L, Jutkowitz E, Lyketsos CG. Reducing neuropsychiatric symptoms in persons with dementia and associated burden in family caregivers using tailored activities: Design and methods of a randomized clinical trial. Contemp Clin Trials. 2016 Jul;49:92-102. doi: 10.1016/j.cct.2016.06.006. Epub 2016 Jun 21. PMID 27339865
- [Derived] Hodgson NA, Gooneratne N, Perez A, Talwar S, Huang L. A timed activity protocol to address sleep-wake disorders in home dwelling persons living with dementia: the healthy patterns clinical trial. BMC Geriatr. 2021 Aug 3;21(1):451. doi: 10.1186/s12877-021-02397-2. PMID 34344312
- [Derived] Hwang Y, Connell LM, Rajpara AR, Hodgson NA. Impact of COVID-19 on Dementia Caregivers and Factors Associated With their Anxiety Symptoms. Am J Alzheimers Dis Other Demen. 2021 Jan-Dec;36:15333175211008768. doi: 10.1177/15333175211008768. PMID 33853394

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Persons living with dementia (PLWDs) and their caregivers (also referred to as dyads) are randomly assigned to either the timed activity intervention or the attention control group. All dyads are screened for eligibility prior to enrollment and randomization. The study enrolled one dyad that is not counted in the enrollment number - they were unable to be randomized after enrollment due to home safety concerns.
Groups:
- Caregivers of Persons Living With Dementia: Timed Activity Intervention Protocol; People Living With Dementia: Timed Activity Intervention Protocol: The timed activity group will be delivered to caregivers and persons living with dementia, and will involve 4 in-home visits and 4 brief telephone education sessions provided over 4 weeks. The timed activity intervention provides activities delivered at specific times in the daily cycle. The in-home sessions are spaced weekly so that the participants can have the opportunity to practice the activity with the interventionist and then on their own. During each session, the interventionist will reinforce activity use, review problem solving approaches, and provide education.
  Timed Activity Intervention: The timed activity group will involve 4 in-home visits and 4 brief telephone education sessions provided over 4 weeks. The timed activity intervention provides activities delivered at specific times in the daily cycle. The in-home sessions are spaced weekly so that the participants can have the opportunity to practice the activity with the interventionist and then on their own. During each session, the interventionist will reinforce activity use, review problem-solving approaches, and provide education.
- Caregivers of Persons Living With Dementia: Attention-Control Condition; Persons Living With Dementia: Attention-Control Condition: The attention control group sessions will be delivered to caregivers and persons living with dementia.
  This condition will contain no active elements beyond its nonspecific components, and no theoretical basis to support an effect on CRDs. The attention-control group will also involve 4 in-home visits and 4 brief telephone education sessions. The attention control group will receive printed educational and training materials from the Alzheimer's Association and the NIH on home modification, health promotion, talking to your doctor, and advanced care planning that coincide with session content.
  Attention-Control Condition: This condition will contain no active elements beyond its nonspecific components, and no theoretical basis to support an effect on CRDs. The attention-control group will also involve 4 in-home visits and 4 brief telephone education sessions. The attention control group will receive printed educational and training materials from the Alzheimer's Association and the NIH on home modification, health promotion, talking to your doctor, and advanced care planning that coincide with session content.
- Unrandomized: Unrandomized Participants who were consented but didn't move forward in the intervention.
Period: Overall Study
Arm/Group | Caregivers of Persons Living With Dementia: Timed Activity Intervention Protocol | Caregivers of Persons Living With Dementia: Attention-Control Condition | People Living With Dementia: Timed Activity Intervention Protocol | Persons Living With Dementia: Attention-Control Condition | Unrandomized
Started | 105 | 105 | 105 | 105 | 1
Completed | 94 | 95 | 94 | 95 | 0
Not Completed | 11 | 10 | 11 | 10 | 1
Not completed — Lost to Follow-up | 4 | 7 | 4 | 7 | 1
Not completed — Withdrawal by Subject | 7 | 3 | 7 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | People Living With Dementia: Timed Activity Intervention Protocol | Persons Living With Dementia: Attention-Control Condition | Caregivers of Persons Living With Dementia: Timed Activity Intervention Protocol | Caregivers of Persons Living With Dementia: Attention-Control Condition | Total
Number analyzed (Participants) | 105 | 105 | 105 | 105 | 420
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Some demographic characteristics missing for two participants.
  years
    number analyzed (Participants) | 104 | 104 | 96 | 95 | 399
    (all) | 73.5 (8.4) | 73.9 (8.9) | 57.5 (14.2) | 55.6 (15.3) | 65.13 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Some demographic characteristics missing for two participants.
  Participants
    number analyzed (Participants) | 104 | 105 | 104 | 105 | 418
    Female | 67 | 72 | 67 | 72 | 278
    Male | 37 | 33 | 37 | 33 | 140
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Some demographic characteristics missing for two participants.
  Participants
    number analyzed (Participants) | 104 | 105 | 104 | 105 | 418
    Hispanic or Latino | 18 | 21 | 18 | 21 | 78
    Not Hispanic or Latino | 85 | 83 | 85 | 83 | 336
    Unknown or Not Reported | 1 | 1 | 1 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 65 | 70 | 64 | 70 | 269
  White | 39 | 34 | 40 | 34 | 147
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 1 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in the Quality of Life in Alzheimer's Disease (QOL-AD) Scale
Description: Person living with dementia quality of life. The QOL-AD scale uses a scale of 1-4 (poor, fair, good, or excellent) to rate a variety of life domains, including the patient's physical health, mood, relationships, activities, and ability to complete tasks. Total scores are calculated by summing all domain scores. The total score range is 13 to 52, with higher scores indicating higher quality of life. Total scores were analyzed to see if there was a change from baseline to one month. The change was calculated from two time points as the value at the later time point minus the value at the earlier time point. Change scores are reported.
Time Frame: Baseline and 1 month
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | People Living With Dementia: Timed Activity Intervention Protocol | Persons Living With Dementia: Attention-Control Condition
Number analyzed (Participants) | 105 | 105
scores on a scale | 0.56 (4.06) | -0.47 (5.16)

2. Secondary Outcome: Neuropsychiatric Inventory (NPI)
Description: Neuropsychiatric Behaviors The Neuropsychiatric Inventory Questionnaire (NPI) is an informant-based instrument that measures the presence and severity of 12 Neuropsychiatric Symptoms (NPS) in patients with dementia, as well as informant distress.
  Neuropsychiatric symptoms are rated by the caregiver within a domain in terms of both frequency (1=rarely, less than once per week; 2=sometimes, about once per week; 3=often, several times per week; and 4=very often, once or more per day) and severity (1=mild; 2=moderate; 3=severe), thus yielding a composite symptom domain score (frequency × severity) ranging from 0 (absence of behavioral symptoms) to 144 points (maximum severity of behavioral symptoms).
Time Frame: 4 Months
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Circadian Rhythm Symptoms From Actigraphy
Description: Measured using a Motionlogger actigraphy bracelet worn by CR for consecutive 24-hour periods for one whole month.
  Actigraphic measures of physical activity do not rely on participant self-report and may be of particular importance for efforts to examine the health benefits of physical activity across the full spectrum of older individuals especially those with dementia, a group in which loss of motor function is particularly salient.
Time Frame: 30 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during time of participant enrollment (one month of active participation, three-month follow-up after completion of study).
Groups:
- Unrandomized: Participants who were not randomized into the study.
Arm/Group | Unrandomized | People Living With Dementia: Timed Activity Intervention Protocol | Persons Living With Dementia: Attention-Control Condition | Caregivers of Persons Living With Dementia: Timed Activity Intervention Protocol | Caregivers of Persons Living With Dementia: Attention-Control Condition
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/105 | 0/105 | 0/105 | 0/105
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/105 | 0/105 | 0/105 | 0/105
Other Adverse Events (participants affected / at risk) | 1/1 | 6/105 | 5/105 | 0/105 | 0/105
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Unrandomized (N=1) | People Living With Dementia: Timed Activity Intervention Protocol (N=105) | Persons Living With Dementia: Attention-Control Condition (N=105) | Caregivers of Persons Living With Dementia: Timed Activity Intervention Protocol (N=105) | Caregivers of Persons Living With Dementia: Attention-Control Condition (N=105)
Hospitalization (Injury, poisoning and procedural complications) | 0 | 2 | 4 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Caregiver agitation (Social circumstances) | 0 | 1 | 0 | 0 | 0
Wandering (Social circumstances) | 0 | 1 | 0 | 0 | 0
Lack of caregiver support (Social circumstances) | 0 | 1 | 0 | 0 | 0
Infestation (Infections and infestations) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-02): https://cdn.clinicaltrials.gov/large-docs/85/NCT03682185/Prot_SAP_000.pdf